CLINICAL TRIAL: NCT00224822
Title: The Effects of Aripiprazole on Patients With "Metabolic Syndrome": An Open-Label Trial
Brief Title: The Effects of Aripiprazole on Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New Mexico VA Healthcare System (U.S. Federal Agency)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA-0001; BRINM #170
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Metabolic Syndrome X
Keywords: Psychiatry; Antipsychotic; Psychopharmacology; Clinical Trial; Open Label; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Metabolic Syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Metabolic Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The primary goal of this study is to assess the effect of aripiprazole on patients who developed metabolic syndrome while taking other second generation antipsychotic medications.

DETAILED DESCRIPTION:
Schizophrenia, schizoaffective disorder and bipolar disorder are severe and disabling disorders, associated with marked social or occupational dysfunction, tenfold suicidal risk, intensive healthcare resource utilization and poor prognosis. Atypical antipsychotics developed in the last decade are proving beneficial to a subset of patients. These agents share a reduced risk for EPS and tardive dyskinesia in comparison with first generation antipsychotics. They also appear to improve negative, cognitive, and depressive symptoms while being at least as efficacious as first generation "typical" drugs in controlling positive symptoms of schizophrenia and schizoaffective disorder. Unfortunately, during the late 1990's, case reports and studies began to document a number of adverse events associated with the use of most second generation antipsychotics such as weight gain, hyperlipidemia and hyperglycemia subsumed under the name "metabolic syndrome". Aripiprazole has a unique pharmacological mechanism, making this drug the ideal medication for treatment to patients who experience metabolic syndrome from other second generation antipsychotics. In numerous pervious trials, it has been demonstrated that aripiprazole is a safe and effective treatment for schizophrenia, schizoaffective disorder and bipolar disorder and that it may actually reduce plasma glucose levels and improve lipid profiles, lowering the risk for cardiovascular disease and /or diabetes. Thirty patients with Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder who have experienced a 10 pound increase in weight while on a second generation antipsychotic or hyperlipidemia, or hyperglycemia, will switch to aripiprazole and be monitored for any improvement in BMI, lipids and glucose.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder who, based on chart review, have developed significant weight gain or any clinically significant aspect of the metabolic syndrome including weight gain, hyperglycemia, diabetes, or hyperlipidemia, while on a second generation antipsychotic medication.
* Between 18-65 years of age
* Decisional capacity is adequate to provide informed consent or has an authorized appropriate surrogate decision maker.
* If female, must agree to use a medically approved contraceptive or does not possess potential to bear children

Exclusion Criteria:

* History of adverse reaction to aripiprazole
* Serious hepatic, renal, cardiac, neurological, or pulmonary disease that would prevent safe participation in a drug trial
* A diagnosis of active drug or alcohol abuse according to DSM-IV criteria within the last 30 days
* Suicidal or homicidal ideation or psychotic decompensation
* Patients on Paxil, Remeron, tricyclic or monoamine oxidase inhibitor (MAOI) antidepressants or mood stabilizers other than lamotrigine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome assessment is weight gain/body mass index (BMI) compared to baseline
Other primary outcomes with regard to efficacy will be scores on the Brief Psychiatric Rating Scale (BPRS) and Clinical Global Impressions (CGI) compared to baseline.

SECONDARY OUTCOMES:
Fasting lipids, glucose profiles and electrocardiogram (EKG) results compared to baseline to assess glucose, weight, lipids, and heart rhythms

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Geppert, MD, PhD, Principal Investigator — New Mexico VA Healthcare System
Locations (1):
- New Mexico VA Healthcare System, Albuquerque, New Mexico, United States

REFERENCES:
- See also: The New Mexico VA Healthcare System website — http://www.albuquerque.va.gov/
- See also: The website for the Biomedical Research Institute of New Mexico — http://www.brinm.org